CLINICAL TRIAL: NCT06716242
Title: Prospective, Observational, Multicentre Study to Confirm the Performance of Molecular Screening for Early Detection of Preeclampsia
Brief Title: Validation of the MaiRa Preeclampsia Test for Screening Early/Late Preeclampsia in First and Second Trimesters
Acronym: iPregnostic
Status: Recruiting | Type: Observational
Sponsor: iPremom (Industry)
Responsible Party: Sponsor
Other Study IDs: IPR-IPR-TG-24-01
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Preeclampsia (PE)
Keywords: Early Screening; First Trimester Diagnostic; Cell-Free RNA (cfRNA); Molecular Profile; Blood Biomarkers
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with cfRNA/DNA and other biomolecules. Maternal peripheral blood samples analyzed for C-RNA, cfRNA, DNA, and other markers linked to preeclampsia and obstetric outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant patients aged 18 years or older: Pregnant patients aged 18 years or older recruited between 9 and 14 weeks' gestation during routine obstetrical follow-ups at referral hospitals.
  Interventions: Procedure: Peripheral blood collection

INTERVENTIONS:
Procedure: Peripheral blood collection — Maternal peripheral blood will be collected 3 times during pregnancy (1st, 2nd and 3rd trimester) and clinical data will also be compiled.

SUMMARY:
Preeclampsia (PE) is a major obstetric complication with severe short- and long-term consequences for both mother and fetus. Early detection is critical to mitigate PE-related morbidity and mortality. Effective screening tools are needed to identify women at risk, enabling timely preventive and therapeutic interventions.

Current screening methods primarily target placental biomarkers like sFLT1 and PlGF, which are limited to short-term predictions near symptom onset. Existing first-trimester assessments that incorporate maternal factors and Doppler metrics remain constrained by low sensitivity (<41%) in compliance with NICE and ACOG guidelines.

Recent advancements in cell free RNA (cf-RNA) analysis have revealed potential in first-trimester PE prediction. Findings from the PREMOM study (NCT04990141) established a molecular profile for early-onset preeclampsia (EOPE) and late-onset preeclampsia (LOPE) through cfRNA analysis, culminating in the development of the MaiRa Preeclampsia Test (Maternal Advanced and Innovative Preeclampsia Risk Assessment), which demonstrated high predictive performance for first- and second-trimester screening.

The current study hypothesizes that the MaiRa Preeclampsia Test is generalizable, maintaining its predictive accuracy in an independent cohort.

DETAILED DESCRIPTION:
This multicentre, prospective observational study aims to validate the MaiRa Preeclampsia Test, a molecular screening tool for predicting early-onset preeclampsia (EOPE) and late-onset preeclampsia (LOPE) in the first and second trimesters of pregnancy. The study will evaluate its diagnostic accuracy, including sensitivity, specificity, predictive values, and area under the curve (AUC).

Study Design:

Duration: 30 months

* Recruitment and Sample Collection: 18 months
* Sample Analysis: 12 months
* Follow-Up: 8 months
* Statistical Analysis and Publication: 6 months Participants: 7,473 pregnant women from 12 tertiary hospitals in Spain.

Visits:

* Visit 1 (T1): 9-14 weeks' gestation (first blood sample)
* Visit 2 (T2): 15-26 weeks' gestation (second blood sample)
* Visit 3 (T3): ≥27 weeks' gestation (third blood sample)

Blood samples will be analyzed using the MaiRa Preeclampsia Test, with results correlated against obstetric outcomes as the gold standard. Data will be documented in an electronic Case Report Form (eCRF). Quality assurance will be maintained via continuous data monitoring and verification.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent approved by the Ethics Committee.
* Women ≥18 years of age at consent.
* Single gestation pregnancies with first sample collection (T1) possible between 9 and 14 weeks' gestation.

Exclusion Criteria:

* Active neoplasm.
* History of organ or bone marrow transplantation.
* Maternal transfusion within 8 weeks before sample collection.
* Evidence of early pregnancy loss at consent.
* Severe, uncontrolled infections.
* Other investigator-assessed risks that could compromise participation or data quality.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant patients aged 18 years or older, recruited between 9 and 14 weeks' gestation during routine obstetrical follow-ups at referral hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 7473 (Estimated)
Dates: Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Validation of the MaiRa Preeclampsia Test for first-trimester screening (9-14 weeks) of EOPE | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks.
  Sensitivity, specificity, accuracy, F1-score, positive/negative predictive values, false discovery rate, AUC.

SECONDARY OUTCOMES:
Validation of second-trimester screening (15-26 weeks) for EOPE | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks.
  Sensitivity, specificity, accuracy, F1-score, positive/negative predictive values, false discovery rate, AUC.
Validation of second-trimester screening (15-26 weeks) for LOPE | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks.
  Sensitivity, specificity, accuracy, F1-score, positive/negative predictive values, false discovery rate, AUC.

OTHER OUTCOMES:
Exploratory outcome: Validation of first-trimester screening (9-14 weeks) for LOPE | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks.
  Sensitivity, specificity, accuracy, F1-score, positive/negative predictive values, false discovery rate, AUC.
Exploratory outcome: Validation of first and second trimester screening for other pregnancy complications | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks.
  Other pregnancy complications such as preterm labour, intrauterine growth restriction, gestational diabetes and placenta previa among others.
  Sensitivity, specificity, accuracy, F1-score, positive/negative predictive values, false discovery rate, AUC.
Exploratory outcome: Molecular characterization of cfRNA and other biomarkers across gestation | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks.
  DNA/RNA/proteins/metabolites associated with gestational age and clinical outcomes.
Exploratory outcome: Identification of candidate biomarkers in maternal blood for therapeutic interventions | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks.
  Molecular characterization (DNA/RNA/proteins/metabolites).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simón, MD, PhD, Principal Investigator — Carlos Simon Foundation; Tamara Garrido, PhD, Principal Investigator — iPremom
Locations (11):
- Spain (11):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Comarcal de Vinaròs, Vinaròs, Castellón
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital de Manises, Manises, Valencia
  - Hospital Universitario Doctor Peset, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia